CLINICAL TRIAL: NCT05541029
Title: Music Listening Interventions for Children Receiving Mechanical Ventilation: A Mechanistic Trial
Brief Title: Music Listening: A Mechanistic Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jessica Jarvis, Postdoctoral Research Fellow, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY22080069; K23HD106011 (NIH)
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Critical Illness
Keywords: mechanical ventilation; pain; stress; anxiety
MeSH Terms: conditions — Critical Illness; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants will receive 3 conditions in a random order, via within-subject block randomization, each day for 3 consecutive days.
Who Masked: Outcomes Assessor
Masking Description: Study team members responsible for collecting data pre-post session will be masked to the condition received and condition order.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Live music > Recorded music > Usual Care (Experimental): Order of conditions for the day
  Interventions: Behavioral: Live music; Behavioral: Recorded music; Other: Usual care
- Recorded music > Usual care > Live music (Experimental): Order of conditions for the day
  Interventions: Behavioral: Live music; Behavioral: Recorded music; Other: Usual care
- Usual Care > Live music > Recorded music (Experimental): Order of conditions for the day
  Interventions: Behavioral: Live music; Behavioral: Recorded music; Other: Usual care
- Live music > Usual Care > Recorded music (Experimental): Order of conditions for the day
  Interventions: Behavioral: Live music; Behavioral: Recorded music; Other: Usual care
- Recorded music > Live music > Usual care (Experimental): Order of conditions for the day
  Interventions: Behavioral: Live music; Behavioral: Recorded music; Other: Usual care
- Usual care > Recorded music > Live music (Experimental): Order of conditions for the day
  Interventions: Behavioral: Live music; Behavioral: Recorded music; Other: Usual care

INTERVENTIONS:
Behavioral: Live music — Live Music. A board-certified music therapist will provide live music (singing with instrument accompaniment) of child preferred songs, per caregiver report, with the tempo entrained to the child's respiratory rate at intervention start and decreased as needed to facilitate relaxation, with a target tempo of 60-80 beats per minute (BPM). Song choices will be based on patient preferences, per caregiver report, and performed with relaxing characteristics (steady rhythm and volume)
Behavioral: Recorded music — Recorded Music. MP3 players will be loaded with a recorded music playlist of the child's preferred songs, per caregiver report, and connected to two small speakers that are to be placed at either side of the head of the bed. Speakers will be tested with sound level meter and volume control set at 50-60 decibels. A member of the study team will stay at bedside throughout the recorded music condition. Study team member will log time of session and complete a checklist with open-response option to note relevant information (e.g., Session interruptions from other staff).
Other: Usual care — Usual Care. A pharmacologic approach to ameliorating stress and pain in MV children is standard of care in CHP's PICU. CHP provides weight-based guidelines to aid clinical decisions on medications for sedation and analgesia. Bedside nurses assess the child's sedation and pain scores once an hour and administered PRN medications as needed, based on clinical judgement, using CHP's PICU weight-based guidelines. For example, if a child has a pain score of >1-2 above goal, guidelines suggest providing a fentanyl dose of 0.5 mcg/kg and assessing again in 1 hour. We will include usual care as a third condition to explore how our selected biomarkers vary over 20 min. without the addition of any musical stimuli. A member of the study team will stay at bedside throughout the usual care condition. Study team member will log time of session and complete a checklist with open-response option to note relevant information (e.g., Session interruptions from other staff).

SUMMARY:
A randomized within-subject crossover trial to compare the effects of live and recorded music listening on biomarkers of stress and pain among children receiving mechanical ventilation in the pediatric intensive care unit.

DETAILED DESCRIPTION:
Children who are critically ill and receiving mechanical ventilation are at increased risks for experiencing high levels of stress and pain, which negatively impacts immediate and long-term health. The current standard of care for treating stress and pain is to provide analgesic and sedative medications, which are associated with increased risk of delirium and posttraumatic stress disorder. This randomized within-subject crossover trial will compare the effects of live and recorded music listening on biomarkers of stress and pain among children receiving mechanical ventilation in the pediatric intensive care unit, to identify the key components of a music listening intervention and explore its mechanism of action, i.e., the biological pathway through which music listening decreases stress and pain.

ELIGIBILITY:
Inclusion Criteria:

* 2 months -17 years old
* intubated and receiving MV
* expected to have a PICU stay of >72 hours

Exclusion Criteria:

* Primary caregiver does not read, write, and speak English
* The child is not expected to survive the PICU stay
* The child has deafness in both ears, has a history of musicogenic epilepsy, is receiving neuromuscular blockade infusion
* The child has a diagnosis of COVID-19
* The child was admitted for a new traumatic brain injury

Ages: 2 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 171 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2027-04-08 (Estimated); Study Completion 2027-05-03 (Estimated)

PRIMARY OUTCOMES:
Change in cortisol pre-post condition | Change from baseline to 30 min. and 60-90 min. post each condition for up to 3 days
  Percent change in saliva-based cortisol level, ng/ml. Reported as median change per condition and included as continuous outcome in linear regression.
Change in Interleukin-6 (IL6) pre-post condition | Change from baseline to 30 min. and 60-90 min. post each condition for up to 3 days
  Percent change in saliva-based IL6 level, pg/ml. Reported as median change per condition and included as continuous outcome in linear regression.
High Frequency (HF) Heart Rate Variability | 1 hour prior through 2 hours post each condition, up to 3 days
  Trajectory of HF, a biomarker of sympathetic nervous activity. Reported as median value per condition and included as continuous outcome in linear regression.
Low Frequency (LF) Heart Rate Variability | 1 hour prior through 2 hours post each condition, up to 3 days
  Trajectory of LF, a biomarker of parasympathetic nervous activity. Reported as median value per condition and included as continuous outcome in linear regression.
HF to LF ration (HF/LF) Heart Rate Variability | 1 hour prior through 2 hours post each condition, up to 3 days
  Trajectory of HF/LF ratio, a biomarker of autonomic nervous system balance. Reported as median value per condition and included as continuous outcome in linear regression.
Standard Deviation of Normal to Normal (SDNN) Heart Rate Variability | 1 hour prior through 2 hours post each condition, up to 3 days
  Trajectory of SDNN, a biomarker of parasympathetic and sympathetic modulation

SECONDARY OUTCOMES:
Acceptability | Interviews conducted within 1 month of completing primary data collection
  Qualitative interviews with participants on intervention benefits, limitations, and optimizations. Reported as themes and sub-themes.
Change in Visual Analogue Scale of Anxiety | Change <30 min. pre-post each condition for up to 3 days
  Percent change in caregiver self-reported anxiety, scaled 0 [no anxiety] to 100 [extremely anxious]. Reported as median change per condition and included as continuous outcome in linear regression.
Change in Face Legs Activity Consolability and Crying (FLACC) | Change <30 min. pre-post each condition for up to 3 days
  Percent change in observed pain, as measured by FLACC. Each of the 5 domains (e.g., Face, legs, etcs) is scored 0-2 and combined for a total score of 0 through 10, higher number indicates more pain. FLACC change score will be calculated from scores pre/post each condition. Reported as median change per condition and included as continuous outcome in linear regression.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica M Jarvis, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chlan LL, Weinert CR, Heiderscheit A, Tracy MF, Skaar DJ, Guttormson JL, Savik K. Effects of patient-directed music intervention on anxiety and sedative exposure in critically ill patients receiving mechanical ventilatory support: a randomized clinical trial. JAMA. 2013 Jun 12;309(22):2335-44. doi: 10.1001/jama.2013.5670. PMID 23689789
- [Background] Liu MH, Zhu LH, Peng JX, Zhang XP, Xiao ZH, Liu QJ, Qiu J, Latour JM. Effect of Personalized Music Intervention in Mechanically Ventilated Children in the PICU: A Pilot Study. Pediatr Crit Care Med. 2020 Jan;21(1):e8-e14. doi: 10.1097/PCC.0000000000002159. PMID 31652195
- [Background] Bush HI, LaGasse AB, Collier EH, Gettis MA, Walson K. Effect of Live Versus Recorded Music on Children Receiving Mechanical Ventilation and Sedation. Am J Crit Care. 2021 Sep 1;30(5):343-349. doi: 10.4037/ajcc2021646. PMID 34467386